CLINICAL TRIAL: NCT07152249
Title: Advancing Strategies to Optimize the PerIopeRativE Management of PostOperative Nausea and Vomiting (ASPIRE-PONV) Trial
Acronym: ASPIRE-PONV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Miklos Kertai, Professor Cardiothoracic Anesthesiology, Vice Chair Perioperative Medicine, Director Perioperative Precision Medicine Program, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 250773
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Nausea; Postoperative Vomiting
Keywords: clinical decision support
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: This trial will use a repeated crossover design. The planned 12-month period of enrollment will be divided into four 12 -week blocks (10 weeks of control or intervention followed by a 2-week washout period).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention will be delivered.
- Anesthesia Workflow-Driven Clinical Decision Support (AW-D CDS) Tool Intervention (Experimental): The AW-D CDS Tool will test the delivery of PONV prophylaxis with the use of the clinical decision support tool. When a patient meets the study study criteria, the AW-D CDS Tool will provide automated notification through the electronic health system.
  The automated notifications be triggered and linked to the point-of-care/desired time of PONV medication administration throughout the workflow of the anesthetic case to optimize the timing of PONV medication administration (pre-procedure evaluation, post-induction, pre-emergence).
  The provider is not forced to follow the recommendations, rather it serves as a reminder of best practices as defined by our department.
  The intervention will be assessed using a repeated cross-over design at the institutional level with periods of time for washout, control and study intervention.
  Interventions: Other: AW-D Clinical Decision Support Tool

INTERVENTIONS:
Other: AW-D Clinical Decision Support Tool — The AW-D Clinical Decision Support Tool will test the automatic delivery of best practice advisories for antiemetic medications at critical timepoints in the perioperative period.
  Arms: Anesthesia Workflow-Driven Clinical Decision Support (AW-D CDS) Tool Intervention

SUMMARY:
The goal of this prospective, unblinded, pragmatic and repeated crossover trial is to learn if clinical decision support alerts will impact postoperative nausea and vomiting (PONV) prophylaxis and reduce PONV rates in adult patients who have planned surgery with general anesthesia. The main aim is to improve PONV, establishing a scalable Clinical Decision Support (CDS) Tool for personalized PONV prevention.

The primary hypothesis is that, compared with standard care, the Anesthesia Workflow-Driven Clinical Decision Support Tool for Personalized PONV Prevention will be associated with a significant improvement in the rate of appropriate administration of PONV prophylaxis and a significant decrease in the incidence of PONV.

This study will evaluate a new clinical decision support (CDS) tool designed to improve how and when PONV prevention strategies are used. Unlike traditional tools that provide generic, one-time alerts, this new system is integrated into the electronic health record (EHR) and delivers timely, targeted reminders to anesthesia providers at key moments during a patient's surgical care-such as before surgery begins, after anesthesia is given, and before the patient wakes up. These alerts are based on each patient's individual risk for PONV and are intended to support, not replace, clinical judgment. The study will use a crossover design over 12 months, alternating between periods when the tool is active and when it is not. The goal is to determine whether this time-sensitive, workflow-integrated tool can lead to better adherence to best practices and improved patient outcomes.

ELIGIBILITY:
Adult Inclusion Criteria

* Age ≥ 18 years
* Planned surgery with general anesthesia with endotracheal intubation or laryngeal mask airway
* Meet zero or more risk factors for PONV ( history of motion sickness or postoperative nausea and vomiting, non-smoker, female sex, duration of inhalation anesthesia greater than 1 hour, undergoing high risk surgical procedure (cholecystectomy, laparoscopy, gynecologic), and perioperative opioid use)

Adult Exclusion Criteria

* ASA 6 including organ procurement,
* Patients anticipated to be transferred directly to the intensive care unit intubated,
* Procedure types:

  * Electroconvulsive therapy,
  * Intubation only cases,
  * labor epidurals,
  * transesophageal echocardiography (TEE)/cardioversion,
  * surgery duration < 30 minutes.

Operating Room Anaesthesia Provider Inclusion Criteria

Any operating room anaesthesia provider of eligible patients will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19480 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Adult patients: rate of appropriate administration of PONV prophylaxis | Intraoperative
  For adult patients (PONV-5), the rate of appropriate administration of PONV prophylaxis based consensus guidelines and standardized institutional protocols. For the definition of the primary outcome we will be using the definition set by the Michigan PeriOperative Group ASPIRE Program, as follows: adult patients with PONV-05, "are ≥18 years old who had a procedure requiring general anesthesia or cesarean delivery and administered appropriate prophylaxis for PONV"

SECONDARY OUTCOMES:
Adult Patients: incidence of PONV | 3 hours postoperatively
  Adult Patients: Incidence of PONV as defined by MPOG ASPIRE: Presence of i) PONV-03b, EHR documented nausea/vomiting in the immediate postoperative period, and/or ii) PONV-03, EHR documented PONV OR rescue antiemetic administration in the immediate postoperative period.
Adult Patients: PACU length of stay | PACU admission to discharge (usually 1-3 hours post operatively)
  Duration of time spent in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Kertai, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stallings EG, Wanderer JP, Balavage M, Henson CP, Fowler L, Eden S, Shotwell MS, Gruss C, Neuhafen KR, Gelfand BJ, Kertai MD; ASPIRE-PONV Investigators. Advancing Strategies to Optimise the PerIopeRativE Management of PostOperative Nausea and Vomiting (ASPIRE-PONV) study: rationale and design for a sequential, repeated crossover trial. BMJ Open. 2026 Feb 10;16(2):e113842. doi: 10.1136/bmjopen-2025-113842. PMID 41667172